CLINICAL TRIAL: NCT04677283
Title: Study of Symptoms Linked to Covid-19 in Residents and Professionals in EHPAD, Associated With a Dual Diagnostic Approach by PCR and Serology: a Cohort in Île-de-France.
Acronym: COVID - EHPAD
Status: Completed | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01027-32
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Symptoms Related to Covid-19
Keywords: Covid-19; serology; Reverse Transcriptase PCR
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose is to study the prevalence of Covid-19 in EHPAD. The primary endpoint will be the combination of PCR results and symptomatology, making it possible to define positive cases in EHPAD, in residents and professionals in contact with them. The prevalence obtained can be compared with the results of serology if these are performed.

DETAILED DESCRIPTION:
This study is taking place in several nursing homes in Ile-de-France, which will be recruited at the end of the diagnostic campaign.

At the initiative of the ARS Ile-de-France, residents and professionals of selected EHPADs will be subjected to systematic screening by RT-PCR for Covid-19, then by serology after the first screening, regardless of whether either the result

Samples, by nasopharyngeal swab for RT-PCR, by capillary blood sampling or venipuncture according to the technique for serology, will be carried out according to the doctrines issued by the ARS Ile de France and the variations proposed by the appropriate departmental directorates in depending on local resources. The results will be brought to the attention of EHPADs to adapt the care of residents and positive professionals.

Data will be collected daily from collection for the first test (RT-PCR), or retrospectively if the collection took place before the study.

Regarding the approach for collecting serologies:

* All subjects included with a negative PCR will be offered the serological test, in accordance with the recommendations in force or the medical decisions of the establishments.
* The qualitative results of the serologies of the subjects included in the study (residents and professionals) will be collected according to the same circuit as those of the RT-PCRs.
* Only the symptoms of residents with a positive serology will be collected, from the date of the sample and for a period of 14 days.
* The symptoms of professionals with a positive serology can be collected, from the date of the sample and for a period of 14 days without mandatory character.
* Both techniques (ELISA or TROD) are accepted and the serology values will not be collected.

ELIGIBILITY:
Inclusion Criteria:

1. / Residents of nursing homes in Île-de-France in which systematic Covid-19 screening tests were carried out and agreeing to participate in the study.
2. / Professionals in nursing homes in Île-de-France in which systematic screening tests for Covid-19 were carried out and agreeing to participate in the study: nursing assistants, nurses, coordinating doctors, hotel and service agents hygiene, etc.

Exclusion Criteria:

1. / Expression of opposition to the collection of symptoms by professionals, residents or their legal representatives.
2. / Subjects who have not had a diagnostic test by RT-PCR.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two types of population, EHPAD residents identified and EHPAD professionals
Sampling Method: Probability Sample
Enrollment: 1059 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
To define positive cases of coronavirus by "Polymerase Chain Reaction" results and symptomatologies | 3 Months

SECONDARY OUTCOMES:
Assessment of commorbidity risk according Charlson score | 3 Months
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 3 Months
Assessment of teh degree of autonomy according AGGIR score | 3 Months
Measuring cognitive impairment according Mini-Mental State Examination (MMSE) scores | 3 Months
Screening for a nutritional disorder according Body Mass Index (BMI) score | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Martine LE NOC - SOUDANI, MD, Study Chair — Autonomy Department; ARS Île-de-France
Locations (1):
- Autonomy Department; ARS Île-de-France, Paris, ARS Île-de-France, France